CLINICAL TRIAL: NCT00258297
Title: A Phase II Safety, Efficacy, and Feasibility Study of Neoadjuvant ZD1839 (IRESSA) in Resectable Esophageal Cancer
Brief Title: Gefitinib in Treating Patients With Stage I, Stage II, or Stage III Esophageal Cancer That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn for lack of funding and accrual
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000447159; URCC-U2203; ZENECA-1839US/0282
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Gefitinib; Neoadjuvant Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gefitinib
Procedure: conventional surgery
Procedure: enzyme inhibitor therapy
Procedure: neoadjuvant therapy
Procedure: protein tyrosine kinase inhibitor therapy
Procedure: surgery

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gefitinib before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well gefitinib works in treating patients with stage I, stage II, or stage III esophageal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of neoadjuvant gefitinib in patients with resectable stage I-III esophageal cancer.

Secondary

* Determine the epidermal growth factor-receptor expression in tissue samples obtained at diagnosis and surgery from patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive oral gefitinib once daily beginning between days -21 and -14 and continuing until day -1. Patients undergo tumor resection on day 0.

After completion of study treatment, patients are followed periodically for 6 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell or adenocarcinoma of the thoracic esophagus

  * Resectable, localized disease with or without metastases in local lymph nodes (T1, T2, or T3; any N; M0)
  * Stage I-III disease
* No known distant metastases
* No cervical-esophageal tumors (upper border < 18 cm from the incisor teeth)
* No supraclavicular metastases

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Adequate bone marrow function

Hepatic

* Adequate hepatic function
* No unstable or uncompensated hepatic disease

Renal

* Creatinine ≤ grade 2 by Common Toxicity Criteria
* Adequate renal function
* No unstable or uncompensated renal disease

Cardiovascular

* No unstable or uncompensated cardiac disease

Pulmonary

* No clinically active interstitial lung disease unless it is asymptomatic with chronic stable radiographic changes
* No unstable or uncompensated respiratory disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known hypersensitivity to gefitinib or any of the excipients
* No other malignancy within the past 2 years except basal cell carcinoma or carcinoma in situ of the cervix
* No evidence of severe or uncontrolled systemic disease
* No other significant clinical disorder or laboratory finding that would preclude study participation

PRIOR CONCURRENT THERAPY:

Endocrine therapy

* Concurrent stable-dose steroids allowed

Surgery

* Recovered from any prior oncologic or other major surgery

Other

* More than 30 days since prior nonapproved or investigational drug
* No prior therapy for this or any other malignancy
* No concurrent phenytoin, carbamazepine, barbiturates, rifampin, or Hypericum perforatum (St. John's wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Effect on the signaling pathways by immunohistochemistry after 2-3 weeks of exposure to gefitinib

CONTACTS AND LOCATIONS:
Overall Officials: Kishan J. Pandya, MD, Study Chair — James P. Wilmot Cancer Center
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States